CLINICAL TRIAL: NCT02746250
Title: Muscle Soreness and Stiffness in Patients With Chronic or Frequent Episodic Tension Type Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lærke Tørring Kolding, Medical student, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-16000619
Record Dates: First submitted 2016-04-13; First posted 2016-04-21 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Tension-type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Amitriptyline; Antidepressive Agents, Tricyclic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tension type headache (Active Comparator): The investigator measures the muscle soreness and muscle stiffness before the patients starts their prescribed treatment with amitriptyline - and again after they have reached their optimal dosage of amitriptyline.
  Interventions: Drug: Amitriptyline
- Healthy controls (No Intervention): The investigator measures the muscle soreness and muscle stiffness once.

INTERVENTIONS:
Drug: Amitriptyline — The investigator recruits patients who have already discussed and agreed to the amitriptyline treatment with their physician. The patients start the treatment after the investigator have measured them once.
  Other Names: Saroten; Tricyclic antidepressants
  Arms: Tension type headache

SUMMARY:
The aim is to investigate muscle soreness and stiffness in patients with Chronic or Frequent Episodic Tension Type Headache before and after treatment with amitriptyline - and to compare the results with healthy individuals.

DETAILED DESCRIPTION:
The muscle stiffness is measured with ultrasonic shear wave elastography in m. masseter, m. sternocleidomastoid and m. Trapezius.

The muscle soreness is measured by palpation of the muscles aided by a so called palpometer.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Tension type headache or frequent episodic tension type headache with at least ten episodes or more per month throughout three months or more.
* Pericranial muscle tenderness

Exclusion Criteria:

* Other primary headache disorder (with the exception of episodic migraine.)
* Pregnancy or ongoing breastfeeding
* Heart disease that contradicts treatment with amitriptyline
* Drug or substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Total Tenderness Score | March 2016 to march 2018. Up to 4 months.
  The soreness of the muscle is reported by the patient on a scale from 0-3 (0= no pain, 1= mild pain, 2= moderate pain and 3= severe pain) when pressure is applied at eight different locations on both sides of the face and neck (m. masseter, m. frontalis, m. pterygoideus lateralis, m. temporalis, m. sternocleidomastoid, pros. mastoideus, m. trapezius and the insertions of the neck muscles at the base of the scull.) The sum of the individual scores make up the total tenderness.
Change in muscle stiffness | March 2016 to march 2018. Up to 4 months.
  The stiffness is measured in terms of the speed of the shear waves (meter/second) the higher the speed the stiffer the muscle.
Change in Local Tenderness Score | March 2016 to march 2018. Up to 4 months.
  Aided by a palpometer a pressure of 160 U is applied to four different locations (m. masseter, m. sternocleidomastoid, the lateral part of m. trapezius and the medial part of the m. trapezius.) At each location the patient report the pain intensity on a scale from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik W Schytz, MD, DMSc, Principal Investigator — Danish Headache Center, Department of neurology, Rigshospitalet Glostrup
Locations (1):
- Danish Headache center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No